CLINICAL TRIAL: NCT02232438
Title: Open Trial of Behavioral Activation Therapy for Depressed or Anxious Adolescents With Cancer
Brief Title: Psychotherapy for Depressed or Anxious Adolescents With Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 6797
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Depression; Anxiety; Cancer
Keywords: Depression; Psychotherapy; Anxiety; Cancer
MeSH Terms: conditions — Depression; Anxiety Disorders; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Behavioral activation therapy (Experimental): Patients treated with Behavioral activation therapy will improve in mood and anxiety symptoms and psychosocial functioning at the end of the 6 weeks of treatment.
  Interventions: Behavioral: Behavioral activation therapy

INTERVENTIONS:
Behavioral: Behavioral activation therapy — Behavioral activation therapy (BAT) is a brief, manualized therapy that has shown efficacy in the treatment of major depressive disorder (MDD) and generalized anxiety disorder (GAD) in several controlled trials patients (see review in Dimidjan et al., Ann Rev Clin Psychol, 2010, and Chu, Brian C., et al. Cognitive and Behavioral Practice, 2009.), including adult cancer patients (Hopkoet al., 2009; Hopko et al., 2011).

SUMMARY:
At present, there are no established treatments for depression or anxiety in adolescents with cancer, creating an important clinical and research gap. Fortunately, there is now substantial evidence documenting the efficacy of psychotherapy in the treatment of depressed and anxious adolescents in the general population.

DETAILED DESCRIPTION:
Despite the high prevalence of depression and anxiety in cancer patients, little is known about the efficacy of psychotherapy in depressed and anxious adolescents with cancer.

Behavioral activation therapy (BAT) is a brief, manualized therapy that has shown efficacy in the treatment of major depressive disorder (MDD) and generalized anxiety disorder (GAD) in several controlled trials patients, including adult cancer patients. The goal of this open label clinical trial is to obtain preliminary evidence of the efficacy of BAT(6 sessions) in a group of adolescent cancer patients with MDD, GAD or adjustment disorder with mood or anxiety features.

We will test the efficacy of BAT using the Multidimensional Anxiety Scale for Children at several time points of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* A primary psychiatric diagnosis of Major Depressive Disorder, Generalized Anxiety Disorder or Adjustment Disorder with Mood or Anxiety features as defined by DSM-IV.
* Cancer patients.
* Parent consent and child assent to participate for patients younger than 18. Patient consent for subjects 18-21.
* Diagnosis of cancer (stage 1-4), but healthy enough to complete study procedures.

Exclusion Criteria:

* Lifetime history of psychosis or bipolar disorder.
* Current suicide risk.
* History of substance abuse or dependence in the three months prior to the study.
* Patients who have ever failed BAT in the context of cancer.
* Receiving other concurrent therapy for same disorder and patients who are receiving effective medication for depression.
* Mental retardation.
* CNS tumors.
* Patients undergoing Stem Cell Transplantation.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in Multidimensional Anxiety Scale for Children (MASC 2) | baseline, and every two weeks till week 10
  10 to 15 minutes of mood assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States